CLINICAL TRIAL: NCT05621148
Title: REfractorinesS to Ibrutinib BTKi and Systemic Targeted Therapy. A FILO Study.
Brief Title: REfractorinesS to Ibrutinib BTKi and Systemic Targeted Therapy
Acronym: RESIST
Status: Completed | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: FILObsLLC_RESIST
Record Dates: First submitted 2022-10-28; First posted 2022-11-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: CLL, Relapsed; CLL, Refractory; Bruton Tyrosine Kinase Inhibitor; Small Lymphocytic Leukemia
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Full population: LLC patients with prior treatment with BTKi - Underlying tenet: these patients have been treated with a BTKi in at least one of two or more prior lines of therapy and progressed - FULL POPULATION
- Narrow population: LLC Patients who progressed BTKi and failed VEN (defined as patients who discontinued VEN due to disease progression, intolerability, or failure to achieve an objective response within 3 months of initiating therapy; small patient population) - Tenet: these patients have been treated with both BTKi and VEN in any one of the prior two lines of therapy and progressed

SUMMARY:
Data evaluating and quantifying real-world outcomes of patients post-ibrutinib discontinuation, as well as outcomes of patients who have progressed on a Bruton tyrosine kinases inhibitors (BTKi) and received prior venetoclax are very limited. There are no robust studies specifically designed to assess outcomes of patients with chronic lymphocytic leukemia (CLL) receiving third line or subsequent treatments. As such, there is no established standard of care for these multiple Relapsed/Refractory (RR) patients. Furthermore, despite new oral agents approved in third-line RR CLL, there are limited published data on how to best sequence these agents and how to manage patients who fail these therapies. As the best salvage therapy in patients who fail all available oral these agents is unknown, this is a population of patients with unmet medical need.

The aim of this study is to determine unmet need and treatment patterns of data from two types of populations, all previously exposed to ibrutinib (or other BTKi) for the full patient population and both ibrutinib (or other BTKi and venetoclax) for the narrow patient population, where these agents failed these subcategories of patient populations, at least in 3rd line therapy (in other words, having at least received two lines of therapy before)

* Patients with prior treatment with BTKi (full patient population) - Underlying tenet: these patients have been treated with a BTKi in at least one of two or more prior lines of therapy and progressed - FULL POPULATION
* Patients who progressed BTKi and failed VEN (defined as patients who discontinued venetoclax (VEN) due to disease progression, intolerability, or failure to achieve an objective response within 3 months of initiating therapy; small patient population) - Tenet: these patients have been treated with both BTKi and VEN in any one of the prior two lines of therapy and progressed. - NARROW POPULATION

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CLL or small lymphocytic leukemia (SLL).
* ≥ 18 years of age the time of initial diagnosis.
* Venetoclax therapy in at least third line of treatment (LOT) during the period considered, following at least one LOT with BTKi
* Patients who received VEN during prior LOTs are eligible.
* Patient not opposed to data collection (including deceased patients)

Exclusion Criteria:

* Exposure to cellular therapy, including CAR T-cells / Allo-Stem Cell Transplantation.
* Richter's transformation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously exposed to ibrutinib (or other BTKi) : treatment with a BTKi in at least one of two or more prior lines of therapy and progressed
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Response rate of treatment patterns in patients with CLL | from BTKi initiation until progression/failure at Venetoclax treatment, assessed up to 7 years
  Overall response rate (complete, partial, stable) for each treatment received

CONTACTS AND LOCATIONS:
Overall Officials: Loïc YSEBAERT, Principal Investigator — French Innovative Leukemia Organisation
Locations (8):
- France (8):
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - Centre Léon Bérard - Hématologie, Lyon
  - Institut Paoli-Calmettes - Hématologie Clinique, Marseille
  - MONTPELLIER - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - Bordeaux Pessac, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse

IPD SHARING:
Plan to Share IPD: No